CLINICAL TRIAL: NCT02622074
Title: A Phase 1b Study to Evaluate Safety and Clinical Activity of Pembrolizumab (MK-3475) in Combination With Chemotherapy as Neoadjuvant Treatment for Triple Negative Breast Cancer (TNBC) - (KEYNOTE 173)
Brief Title: Safety and Efficacy Study of Pembrolizumab (MK-3475) in Combination With Chemotherapy as Neoadjuvant Treatment for Participants With Triple Negative Breast Cancer (TNBC) (MK-3475-173/KEYNOTE-173)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-173; 2015-002405-11 (EudraCT Number); MK-3475-173 (Other: Merck); KEYNOTE-173 (Other: Merck)
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Results first posted 2019-10-24 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-08

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; 130-nm albumin-bound paclitaxel; Anthracyclines; Doxorubicin; Cyclophosphamide; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort A: KNp / KAC (Experimental): Participants receive pembrolizumab (K) 200 mg on Cycle 1 Day 1 followed by pembrolizumab 200 mg in Cycles 2-5 on Day 1 (once every 3 weeks; Q3W) PLUS nab-paclitaxel (KNp) starting at 125 mg/m^2 in Cycles 2-5 on Days 1, 8 and 15 (once each week; QW). This will be followed by pembrolizumab (K) 200 mg in Cycles 6-9 on Day 1 (Q3W) PLUS doxorubicin (A) 60 mg/m^2 in Cycles 6-9 on Day 1 (Q3W) PLUS cyclophosphamide (C) 600 mg/m^2 in Cycles 6-9 on Day 1 (Q3W). All treatments will be administered via intravenous (IV) infusion except for doxorubicin (A), which will be administered via IV injection. Each cycle is 21 days.
  Interventions: Biological: Pembrolizumab; Drug: Nab-paclitaxel; Drug: Anthracycline (doxorubicin); Drug: Cyclophosphamide
- Cohort B: KNpCb (Regimen 1) / KAC (Experimental): Participants first receive KNpCb Regimen 1 which consists of: pembrolizumab (K) 200 mg on Cycle 1 Day 1 PLUS nab-paclitaxel (KNp) starting at 100 mg/m^2 in Cycles 2-5 on Days 1, 8 and 15 (QW) PLUS carboplatin (Cb) starting at Area Under the Curve (AUC) 6 in Cycles 2-5 on Day 1 (Q3W). This will be followed by pembrolizumab (K) 200 mg in Cycles 6-9 on Day 1 (Q3W) PLUS doxorubicin (A) 60 mg/m^2 in Cycles 6-9 on Day 1 (Q3W) PLUS cyclophosphamide (C) 600 mg/m^2 in Cycles 6-9 on Day 1 (Q3W). All treatments will be administered via IV infusion except for doxorubicin (A), which will be administered via IV injection. Each cycle is 21 days.
  Interventions: Biological: Pembrolizumab; Drug: Nab-paclitaxel; Drug: Anthracycline (doxorubicin); Drug: Cyclophosphamide; Drug: Carboplatin
- Cohort C: KNpCb (Regimen 2) / KAC (Experimental): Participants first receive KNpCb Regimen 2 which consists of: pembrolizumab (K) 200 mg on Cycle 1 Day 1 PLUS nab-paclitaxel (KNp) starting at 125 mg/m^2 in Cycles 2-5 on Days 1, 8 and 15 (QW) PLUS carboplatin (Cb) starting at AUC 5 in Cycles 2-5 on Day 1 (Q3W). This will be followed by pembrolizumab (K) 200 mg in Cycles 6-9 on Day 1 (Q3W) PLUS doxorubicin (A) 60 mg/m^2 in Cycles 6-9 on Day 1 (Q3W) PLUS cyclophosphamide (C) 600 mg/m^2 in Cycles 6-9 on Day 1 (Q3W). All treatments will be administered via IV infusion except for doxorubicin (A), which will be administered via IV injection. Each cycle is 21 days.
  Interventions: Biological: Pembrolizumab; Drug: Nab-paclitaxel; Drug: Anthracycline (doxorubicin); Drug: Cyclophosphamide; Drug: Carboplatin
- Cohort D: KNpCb (Regimen 3) / KAC (Experimental): Participants first receive KNpCb Regimen 3 which consists of: pembrolizumab (K) 200 mg on Cycle 1 Day 1 PLUS nab-paclitaxel (KNp) starting at 125 mg/m^2 in Cycles 2-5 on Days 1, 8 and 15 (QW) PLUS carboplatin (Cb) starting at AUC 2 in Cycles 2-5 on Days 1, 8 and 15 (QW). This will be followed by pembrolizumab (K) 200 mg in Cycles 6-9 on Day 1 PLUS doxorubicin (A) 60 mg/m^2 in Cycles 6-9 on Day 1 (Q3W) PLUS cyclophosphamide (C) 600 mg/m^2 in Cycles 6-9 on Day 1 (Q3W) in Cycles 6-9 on Day 1 (Q3W). All treatments will be administered via IV infusion except for doxorubicin (A), which will be administered via IV injection. Each cycle is 21 days.
  Interventions: Biological: Pembrolizumab; Drug: Nab-paclitaxel; Drug: Anthracycline (doxorubicin); Drug: Cyclophosphamide; Drug: Carboplatin
- Cohort E: KTCb (Regimen 1) / KAC (Experimental): Participants first receive KTCb Regimen 1 which consists of: pembrolizumab (K) 200 mg on Cycle 1 Day 1 PLUS paclitaxel (T) starting at 80mg/m^2 in Cycles 2-5 on Days 1, 8, and 15 (QW) PLUS carboplatin (Cb) starting at AUC 5 in Cycles 2-5 on Day 1 (Q3W). This will be followed by pembrolizumab (K) 200 mg in Cycles 6-9 on Day 1 (Q3W) PLUS doxorubicin (A) 60 mg/m^2 in Cycles 6-9 on Day 1 (Q3W) PLUS cyclophosphamide (C) 600 mg/m^2 in Cycles 6-9 on Day 1 (Q3W). All treatments will be administered via IV infusion except for doxorubicin (A), which will be administered via IV injection. Each cycle is 21 days.
  Interventions: Biological: Pembrolizumab; Drug: Anthracycline (doxorubicin); Drug: Cyclophosphamide; Drug: Carboplatin; Drug: Paclitaxel
- Cohort F: KTCb (Regimen 2) / KAC (Experimental): Participants first receive KTCb Regimen 2 which consists of: pembrolizumab (K) 200 mg on Cycle 1 Day 1 PLUS paclitaxel (T) starting at 80mg/m^2 in Cycles 2-5 on Days 1, 8, and 15 PLUS carboplatin (Cb) starting at AUC 2 in Cycles 2-5 on Days 1, 8 and 15 (QW). This will be followed by pembrolizumab (K) 200 mg in Cycles 6-9 on Day 1 (Q3W) PLUS doxorubicin (A) 60 mg/m^2 in Cycles 6-9 on Day 1 (Q3W) PLUS cyclophosphamide (C) 600 mg/m^2 in Cycles 6-9 on Day 1 (Q3W). All treatments will be administered via IV infusion except for doxorubicin (A), which will be administered via IV injection. Each cycle is 21 days.
  Interventions: Biological: Pembrolizumab; Drug: Anthracycline (doxorubicin); Drug: Cyclophosphamide; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Biological: Pembrolizumab — 200 mg administered Q3W as an IV infusion.
  Other Names: MK-3475; KEYTRUDA®
Drug: Nab-paclitaxel — 125 mg/m^2 or 100 mg/m^2 administered weekly as an IV infusion, according to allocation.
  Arms: Cohort A: KNp / KAC; Cohort B: KNpCb (Regimen 1) / KAC; Cohort C: KNpCb (Regimen 2) / KAC; Cohort D: KNpCb (Regimen 3) / KAC
Drug: Anthracycline (doxorubicin) — 60 mg/m^2 administered Q3W as an IV injection.
Drug: Cyclophosphamide — 600 mg/m^2 administered Q3W as an IV infusion.
Drug: Carboplatin — AUC 6 or AUC5 administered Q3W as an IV infusion, or AUC2 administered weekly as an IV infusion, according to allocation.
  Arms: Cohort B: KNpCb (Regimen 1) / KAC; Cohort C: KNpCb (Regimen 2) / KAC; Cohort D: KNpCb (Regimen 3) / KAC; Cohort E: KTCb (Regimen 1) / KAC; Cohort F: KTCb (Regimen 2) / KAC
Drug: Paclitaxel — 80 mg/m^2 or 70 mg/m^2 administered weekly as an IV infusion, according to allocation.
  Arms: Cohort E: KTCb (Regimen 1) / KAC; Cohort F: KTCb (Regimen 2) / KAC

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and clinical activity of pembrolizumab (MK-3475) in combination with six chemotherapy regimens as neoadjuvant treatment for participants with triple negative breast cancer (TNBC).

ELIGIBILITY:
Inclusion Criteria:

* Has previously untreated, locally advanced TNBC.
* Is able to provide 2 core needle biopsies from the primary tumor at screening to the central laboratory and agrees to have a core needle biopsy after single dose pembrolizumab treatment if tumor biopsy is feasible as judged by the investigator.
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has adequate organ function.
* Females of childbearing potential must be willing to use adequate contraception for the course of the study through 12 months after the last dose of study drug for participants receiving cyclophosphamide and through 6 months after the last dose of study drug for participants who do not receive cyclophosphamide.

Exclusion Criteria:

* Has evidence of metastatic breast cancer, concurrent bilateral invasive breast cancer, or inflammatory breast cancer.
* Has another malignancy within the last 5 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative surgery, or in situ cervical cancer.
* Has received prior chemotherapy, targeted therapy, radiation therapy, immunotherapy that targets immune checkpoints, co-stimulatory or co-inhibitory pathways for T cell receptors within the past 12 months.
* Is currently participating and receiving study therapy, or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study drug.
* Has received a live vaccine within 30 days of the first dose of study drug.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B or Hepatitis C.
* Has evidence of current pneumonitis.
* Has a history of non-infectious pneumonitis requiring treatment with steroids or a history of interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has significant cardiovascular disease, such as: History of myocardial infarction, acute coronary syndrome or coronary angioplasty/stenting/bypass grafting within the last 6 months; Congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV or history of CHF NYHA class III or IV
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the study, starting with the screening visit through 12 months after the last dose of trial treatment for participants who have received cyclophosphamide, and for six months after the last dose of study medication for participants who have not.
* Has a known hypersensitivity to the components of the study drug or its analogs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Schmid P, Salgado R, Park YH, Munoz-Couselo E, Kim SB, Sohn J, Im SA, Foukakis T, Kuemmel S, Dent R, Yin L, Wang A, Tryfonidis K, Karantza V, Cortes J, Loi S. Pembrolizumab plus chemotherapy as neoadjuvant treatment of high-risk, early-stage triple-negative breast cancer: results from the phase 1b open-label, multicohort KEYNOTE-173 study. Ann Oncol. 2020 May;31(5):569-581. doi: 10.1016/j.annonc.2020.01.072. Epub 2020 Feb 14. PMID 32278621
- [Derived] Dent R, Cortes J, Park YH, Munoz-Couselo E, Kim SB, Sohn J, Im SA, Holgado E, Foukakis T, Kummel S, Yearley J, Wang A, Nebozhyn M, Huang L, Cristescu R, Jelinic P, Karantza V, Schmid P. Molecular determinants of response to neoadjuvant pembrolizumab plus chemotherapy in patients with high-risk, early-stage, triple-negative breast cancer: exploratory analysis of the open-label, multicohort phase 1b KEYNOTE-173 study. Breast Cancer Res. 2025 Mar 11;27(1):35. doi: 10.1186/s13058-024-01946-y. PMID 40069763
- [Derived] Perez-Garcia J, Soberino J, Racca F, Gion M, Stradella A, Cortes J. Atezolizumab in the treatment of metastatic triple-negative breast cancer. Expert Opin Biol Ther. 2020 Sep;20(9):981-989. doi: 10.1080/14712598.2020.1769063. Epub 2020 May 25. PMID 32450725
- See also: Merck Oncology Clinical Trial Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty participants were allocated and treated on study.
Groups:
- Cohort A: KNp / KAC: Participants received pembrolizumab (K) 200 mg on Cycle 1 Day 1 followed by pembrolizumab 200 mg in Cycles 2-5 on Day 1 (once every 3 weeks; Q3W) PLUS nab-paclitaxel (KNp) starting at 125 mg/m^2 in Cycles 2-5 on Days 1, 8 and 15 (once each week; QW). This was followed by pembrolizumab (K) 200 mg in Cycles 6-9 on Day 1 (Q3W) PLUS doxorubicin (A) 60 mg/m^2 in Cycles 6-9 on Day 1 (Q3W) PLUS cyclophosphamide (C) 600 mg/m^2 in Cycles 6-9 on Day 1 (Q3W). All treatments were administered via intravenous (IV) infusion except for doxorubicin (A), which was administered via IV injection. Each cycle was 21 days.
- Cohort B: KNpCb (Regimen 1) / KAC: Participants first received KNpCb Regimen 1 which consisted of: pembrolizumab (K) 200 mg on Cycle 1 Day 1 PLUS nab-paclitaxel (KNp) starting at 100 mg/m^2 in Cycles 2-5 on Days 1, 8 and 15 (QW) PLUS carboplatin (Cb) starting at Area Under the Curve (AUC) 6 in Cycles 2-5 on Day 1 (Q3W). This was followed by pembrolizumab (K) 200 mg in Cycles 6-9 on Day 1 (Q3W) PLUS doxorubicin (A) 60 mg/m^2 in Cycles 6-9 on Day 1 (Q3W) PLUS cyclophosphamide (C) 600 mg/m^2 in Cycles 6-9 on Day 1 (Q3W). All treatments were administered via IV infusion except for doxorubicin (A), which was administered via IV injection. Each cycle was 21 days.
- Cohort C: KNpCb (Regimen 2) / KAC: Participants first received KNpCb Regimen 2 which consisted of: pembrolizumab (K) 200 mg on Cycle 1 Day 1 PLUS nab-paclitaxel (KNp) starting at 125 mg/m^2 in Cycles 2-5 on Days 1, 8 and 15 (QW) PLUS carboplatin (Cb) starting at AUC 5 in Cycles 2-5 on Day 1 (Q3W). This was followed by pembrolizumab (K) 200 mg in Cycles 6-9 on Day 1 (Q3W) PLUS doxorubicin (A) 60 mg/m^2 in Cycles 6-9 on Day 1 (Q3W) PLUS cyclophosphamide (C) 600 mg/m^2 in Cycles 6-9 on Day 1 (Q3W). All treatments were administered via IV infusion except for doxorubicin (A), which was administered via IV injection. Each cycle was 21 days.
- Cohort D: KNpCb (Regimen 3) / KAC: Participants first received KNpCb Regimen 3 which consisted of: pembrolizumab (K) 200 mg on Cycle 1 Day 1 PLUS nab-paclitaxel (KNp) starting at 125 mg/m^2 in Cycles 2-5 on Days 1, 8 and 15 (QW) PLUS carboplatin (Cb) starting at AUC 2 in Cycles 2-5 on Days 1, 8 and 15 (QW). This was followed by pembrolizumab (K) 200 mg in Cycles 6-9 on Day 1 PLUS doxorubicin (A) 60 mg/m^2 in Cycles 6-9 on Day 1 (Q3W) PLUS cyclophosphamide (C) 600 mg/m^2 in Cycles 6-9 on Day 1 (Q3W) in Cycles 6-9 on Day 1 (Q3W). All treatments were administered via IV infusion except for doxorubicin (A), which was administered via IV injection. Each cycle was 21 days.
- Cohort E: KTCb (Regimen 1) / KAC: Participants first received KTCb Regimen 1 which consisted of: pembrolizumab (K) 200 mg on Cycle 1 Day 1 PLUS paclitaxel (T) starting at 80mg/m^2 in Cycles 2-5 on Days 1, 8, and 15 (QW) PLUS carboplatin (Cb) starting at AUC 5 in Cycles 2-5 on Day 1 (Q3W). This was followed by pembrolizumab (K) 200 mg in Cycles 6-9 on Day 1 (Q3W) PLUS doxorubicin (A) 60 mg/m^2 in Cycles 6-9 on Day 1 (Q3W) PLUS cyclophosphamide (C) 600 mg/m^2 in Cycles 6-9 on Day 1 (Q3W). All treatments were administered via IV infusion except for doxorubicin (A), which was administered via IV injection. Each cycle was 21 days.
- Cohort F: KTCb (Regimen 2) / KAC: Participants first received KTCb Regimen 2 which consisted of: pembrolizumab (K) 200 mg on Cycle 1 Day 1 PLUS paclitaxel (T) starting at 80mg/m^2 in Cycles 2-5 on Days 1, 8, and 15 PLUS carboplatin (Cb) starting at AUC 2 in Cycles 2-5 on Days 1, 8 and 15 (QW). This was followed by pembrolizumab (K) 200 mg in Cycles 6-9 on Day 1 (Q3W) PLUS doxorubicin (A) 60 mg/m^2 in Cycles 6-9 on Day 1 (Q3W) PLUS cyclophosphamide (C) 600 mg/m^2 in Cycles 6-9 on Day 1 (Q3W). All treatments were administered via IV infusion except for doxorubicin (A), which was administered via IV injection. Each cycle was 21 days.
Period: Overall Study
Arm/Group | Cohort A: KNp / KAC | Cohort B: KNpCb (Regimen 1) / KAC | Cohort C: KNpCb (Regimen 2) / KAC | Cohort D: KNpCb (Regimen 3) / KAC | Cohort E: KTCb (Regimen 1) / KAC | Cohort F: KTCb (Regimen 2) / KAC
Started | 10 | 10 | 10 | 10 | 10 | 10
Completed | 6 | 9 | 10 | 9 | 9 | 10
Not Completed | 4 | 1 | 0 | 1 | 1 | 0
Not completed — Death | 4 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: KNp / KAC | Cohort B: KNpCb (Regimen 1) / KAC | Cohort C: KNpCb (Regimen 2) / KAC | Cohort D: KNpCb (Regimen 3) / KAC | Cohort E: KTCb (Regimen 1) / KAC | Cohort F: KTCb (Regimen 2) / KAC | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.5 (11.1) | 49.5 (11.3) | 43.2 (6.4) | 42.3 (11.2) | 56.7 (11.9) | 52.1 (11.3) | 49.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 10 | 10 | 10 | 60
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 10 | 8 | 9 | 10 | 10 | 10 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 2 | 5 | 7 | 1 | 1 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 5 | 8 | 5 | 3 | 9 | 9 | 39
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) Graded Using National Cancer Institute Common Toxicity Criteria for Adverse Events Version 4.0 (NCI CTCAE v4.0)
Description: The following events, if considered to be study-treatment-related by the Investigator, were considered a DLT:
  * Hematologic:
  * Grade 4 neutropenia lasting ≥8 days;
  * Febrile neutropenia Grade 3 or Grade 4; or
  * Grade 4 thrombocytopenia requiring platelet transfusion, or Grade 3 thrombocytopenia with bleeding
  * Non-hematologic:
  * Grade 4 toxicity;
  * Grade ≥3 symptomatic hepatic toxicities lasting >48 hours, or Grade ≥3 asymptomatic hepatic toxicities lasting ≥7 days; or
  * Grade ≥3 non-hematologic, non-hepatic organ toxicity, with exceptions
  * Other:
  * Any treatment delays for ≥14 days due to unresolved toxicity;
  * Grade 5 treatment-related adverse event (AE);
  * A dose reduction of study treatment during the DLT evaluation period.
Time Frame: Cycle 1 Day 1 through end of Cycle 3 and Cycle 6 Day 1 through end of Cycle 7 (Up to ~150 days from first dose of first combination regimen); Each cycle was 21 days.
Population: The DLT evaluable population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: KNp / KAC | Cohort B: KNpCb (Regimen 1) / KAC | Cohort C: KNpCb (Regimen 2) / KAC | Cohort D: KNpCb (Regimen 3) / KAC | Cohort E: KTCb (Regimen 1) / KAC | Cohort F: KTCb (Regimen 2) / KAC
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Participants | 2 | 4 | 6 | 6 | 0 | 4

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment and which does not necessarily have to have a causal relationship with this treatment. The number of participants who experienced an AE either prior to or after definitive surgery is presented.
Time Frame: Up to approximately 28 months (through Interim database cut-off date of 31-May-2018)
Population: The safety population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: KNp / KAC | Cohort B: KNpCb (Regimen 1) / KAC | Cohort C: KNpCb (Regimen 2) / KAC | Cohort D: KNpCb (Regimen 3) / KAC | Cohort E: KTCb (Regimen 1) / KAC | Cohort F: KTCb (Regimen 2) / KAC
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Participants | 10 | 10 | 10 | 10 | 10 | 10

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment and which does not necessarily have to have a causal relationship with this treatment. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 28 months (through Interim database cut-off date of 31-May-2018)
Population: The safety population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: KNp / KAC | Cohort B: KNpCb (Regimen 1) / KAC | Cohort C: KNpCb (Regimen 2) / KAC | Cohort D: KNpCb (Regimen 3) / KAC | Cohort E: KTCb (Regimen 1) / KAC | Cohort F: KTCb (Regimen 2) / KAC
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Participants | 1 | 2 | 1 | 5 | 2 | 5

4. Secondary Outcome: Pathological Complete Response (pCR) Rate Using the Definition of ypT0 ypN0 (No Invasive or Noninvasive Residual in Breast or Nodes)
Description: pCR rate (ypT0 ypN0; no invasive or noninvasive residual in breast or nodes) was defined as the rate of absence of residual invasive and in situ cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by American Joint Committee on Cancer (AJCC) staging criteria assessed by local pathologist at the time of definitive surgery. The percentage of participants with a pCR using the definition of ypT0 ypN0 is presented.
Time Frame: Up to approximately 9 months (at the time of definitive surgery)
Population: The efficacy population consisted of all participants with Baseline evaluable disease by Investigator assessment who started with the recommended Phase 2 dose, regardless of dose modification during the course of the study.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: KNp / KAC | Cohort B: KNpCb (Regimen 1) / KAC | Cohort C: KNpCb (Regimen 2) / KAC | Cohort D: KNpCb (Regimen 3) / KAC | Cohort E: KTCb (Regimen 1) / KAC | Cohort F: KTCb (Regimen 2) / KAC
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Percentage of Participants | 50.0 [22.2 to 77.8] | 80.0 [49.3 to 96.3] | 80.0 [49.3 to 96.3] | 60.0 [30.4 to 85.0] | 20.0 [3.7 to 50.7] | 50.0 [22.2 to 77.8]

5. Secondary Outcome: Pathological Complete Response (pCR) Rate Using the Definition of ypT0/Tis ypN0 (No Invasive Residual in Breast or Nodes; Noninvasive Breast Residuals Allowed)
Description: pCR rate (ypT0/Tis ypN0; no invasive residual in breast or nodes; noninvasive breast residuals allowed) was defined as the rate of absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by AJCC staging criteria assessed by local pathologist at the time of definitive surgery. The percentage of participants with a pCR using the alternative definition of ypT0/Tis ypN0 is presented.
Time Frame: Up to approximately 9 months (at the time of definitive surgery)
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: KNp / KAC | Cohort B: KNpCb (Regimen 1) / KAC | Cohort C: KNpCb (Regimen 2) / KAC | Cohort D: KNpCb (Regimen 3) / KAC | Cohort E: KTCb (Regimen 1) / KAC | Cohort F: KTCb (Regimen 2) / KAC
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Percentage of Participants | 60.0 [30.4 to 85.0] | 80.0 [49.3 to 96.3] | 80.0 [49.3 to 96.3] | 60.0 [30.4 to 85.0] | 30.0 [8.7 to 60.7] | 50.0 [22.2 to 77.8]

6. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Investigator Review: First Combination Regimen
Description: ORR was defined as the percentage of participants who achieved a complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters [SOD] of target lesions) according to RECIST 1.1 by Investigator review. Because imaging was assessed prior to surgery, a confirmation assessment of CR or PR was not obtained. Participants with missing outcome for objective response were considered non-responders. The percentage of participants who experienced a CR or PR based on RECIST 1.1 following the first combination regimen is presented.
Time Frame: At the end of Cycle 5 following treatment with the first combination regimen (KNp, KNpCb, or KTCb) (Up to ~4 months); Each cycle was 21 days.
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: KNp / KAC | Cohort B: KNpCb (Regimen 1) / KAC | Cohort C: KNpCb (Regimen 2) / KAC | Cohort D: KNpCb (Regimen 3) / KAC | Cohort E: KTCb (Regimen 1) / KAC | Cohort F: KTCb (Regimen 2) / KAC
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Percentage of Participants | 60.0 [30.4 to 85.0] | 90.0 [60.6 to 99.5] | 90.0 [60.6 to 99.5] | 90.0 [60.6 to 99.5] | 60.0 [30.4 to 85.0] | 80.0 [49.3 to 96.3]

7. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Investigator Review: Second Combination Regimen
Description: ORR was defined as the percentage of participants who achieved a complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters [SOD] of target lesions) according to RECIST 1.1 by Investigator review. Because imaging was assessed prior to surgery, a confirmation assessment of CR or PR was not obtained. Participants with missing outcome for objective response were considered non-responders. The percentage of participants who experienced a CR or PR based on RECIST 1.1 following the second combination regimen is presented.
Time Frame: After completion of the second combination regimen (KAC; Cycle 9) but prior to surgery (Up to ~9 months); Each cycle was 21 days.
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: KNp / KAC | Cohort B: KNpCb (Regimen 1) / KAC | Cohort C: KNpCb (Regimen 2) / KAC | Cohort D: KNpCb (Regimen 3) / KAC | Cohort E: KTCb (Regimen 1) / KAC | Cohort F: KTCb (Regimen 2) / KAC
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Percentage of Participants | 80.0 [49.3 to 96.3] | 100 [74.1 to 100.0] | 100 [74.1 to 100.0] | 90.0 [60.6 to 99.5] | 70.0 [39.3 to 91.3] | 90.0 [60.6 to 99.5]

8. Secondary Outcome: Event-Free Survival (EFS) Rate at Month 6
Description: EFS was defined as the time from the first dose date of study treatment to any of the following events: progression of disease that precludes definitive surgery, disease recurrence (for participants with complete surgical resection), progression (for participants with incomplete surgical resection), or death due to any cause. Participants without documented events were censored at the date of the last disease status assessment. The Kaplan-Meier estimates of the percentage of participants who were event free at Month 6 are presented (through Final Analysis cut-off of 18-Nov-2019).
Time Frame: Month 6
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: KNp / KAC | Cohort B: KNpCb (Regimen 1) / KAC | Cohort C: KNpCb (Regimen 2) / KAC | Cohort D: KNpCb (Regimen 3) / KAC | Cohort E: KTCb (Regimen 1) / KAC | Cohort F: KTCb (Regimen 2) / KAC
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Percentage of Participants | 90.0 [57.9 to 98.0] | 100.0 [100.0 to 100.0] | 100.00 [100.0 to 100.0] | 90.0 [57.9 to 98.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

9. Secondary Outcome: Event-Free Survival (EFS) Rate at Month 12
Description: EFS was defined as the time from the first dose date of study treatment to any of the following events: progression of disease that precludes definitive surgery, disease recurrence (for participants with complete surgical resection), progression (for participants with incomplete surgical resection), or death due to any cause. Participants without documented events were censored at the date of the last disease status assessment. The Kaplan-Meier estimates of the percentage of participants who were event free at Month 12 are presented (through Final Analysis cut-off of 18-Nov-2019).
Time Frame: Month 12
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: KNp / KAC | Cohort B: KNpCb (Regimen 1) / KAC | Cohort C: KNpCb (Regimen 2) / KAC | Cohort D: KNpCb (Regimen 3) / KAC | Cohort E: KTCb (Regimen 1) / KAC | Cohort F: KTCb (Regimen 2) / KAC
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Percentage of Participants | 80.0 [48.9 to 93.3] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 90.0 [57.9 to 98.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

10. Secondary Outcome: Event-Free Survival (EFS) Rate at Month 24
Description: EFS was defined as the time from the first dose date of study treatment to any of the following events: progression of disease that precludes definitive surgery, disease recurrence (for participants with complete surgical resection), progression (for participants with incomplete surgical resection), or death due to any cause. Participants without documented events were censored at the date of the last disease status assessment. The Kaplan-Meier estimates of the percentage of participants who were event free at Month 24 are presented (through Final Analysis cut-off of 18-Nov-2019).
Time Frame: Month 24
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: KNp / KAC | Cohort B: KNpCb (Regimen 1) / KAC | Cohort C: KNpCb (Regimen 2) / KAC | Cohort D: KNpCb (Regimen 3) / KAC | Cohort E: KTCb (Regimen 1) / KAC | Cohort F: KTCb (Regimen 2) / KAC
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Percentage of Participants | 60.0 [30.9 to 80.1] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 90.0 [57.9 to 98.0] | 90.0 [57.9 to 98.0] | 100.0 [100.0 to 100.0]

11. Secondary Outcome: Overall Survival (OS) Rate at Month 6
Description: OS was defined as the time from the first dose date of study treatment to death due to any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow-up. The Kaplan-Meier estimates of the percentage of participants who were surviving at Month 6 are presented (through Final Analysis cut-off of 18-Nov-2019).
Time Frame: Month 6
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: KNp / KAC | Cohort B: KNpCb (Regimen 1) / KAC | Cohort C: KNpCb (Regimen 2) / KAC | Cohort D: KNpCb (Regimen 3) / KAC | Cohort E: KTCb (Regimen 1) / KAC | Cohort F: KTCb (Regimen 2) / KAC
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Percentage of Participants | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 90.0 [57.9 to 98.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

12. Secondary Outcome: Overall Survival (OS) Rate at Month 12
Description: OS was defined as the time from the first dose date of study treatment to death due to any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow-up. The Kaplan-Meier estimates of the percentage of participants who were surviving at Month 12 are presented (through Final Analysis cut-off of 18-Nov-2019).
Time Frame: Month 12
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: KNp / KAC | Cohort B: KNpCb (Regimen 1) / KAC | Cohort C: KNpCb (Regimen 2) / KAC | Cohort D: KNpCb (Regimen 3) / KAC | Cohort E: KTCb (Regimen 1) / KAC | Cohort F: KTCb (Regimen 2) / KAC
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Percentage of Participants | 80.0 [48.9 to 93.3] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 90.0 [57.9 to 98.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

13. Secondary Outcome: Overall Survival (OS) Rate at Month 24
Description: OS was defined as the time from the first dose date of study treatment to death due to any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow-up. The Kaplan-Meier estimates of the percentage of participants who were surviving at Month 24 are presented (through Final Analysis cut-off of 18-Nov-2019).
Time Frame: Month 24
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: KNp / KAC | Cohort B: KNpCb (Regimen 1) / KAC | Cohort C: KNpCb (Regimen 2) / KAC | Cohort D: KNpCb (Regimen 3) / KAC | Cohort E: KTCb (Regimen 1) / KAC | Cohort F: KTCb (Regimen 2) / KAC
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Percentage of Participants | 70.0 [39.6 to 87.2] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 90.0 [57.9 to 98.0] | 90.0 [57.9 to 98.0] | 100.0 [100.0 to 100.0]

ADVERSE EVENTS:
Time Frame: Up to approximately 45 months (through Final Analysis cut-off date of 18-Nov-2019)
Description: All-Cause Mortality table includes all randomized participants.
  Serious and Other AEs include all randomized participants who received ≥1 dose of study drug. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug were excluded as AEs.
Groups:
- Cohort B: KNpCb (Regimen 1) / KAC: Participants first received KNpCb Regimen 1 which consisted of: pembrolizumab (K) 200 mg on Cycle 1 Day 1 PLUS nab-paclitaxel (KNp) starting at 100 mg/m^2 in Cycles 2-5 on Days 1, 8 and 15 (QW) PLUS carboplatin (Cb) starting at AUC 6 in Cycles 2-5 on Day 1 (Q3W). This was followed by pembrolizumab (K) 200 mg in Cycles 6-9 on Day 1 (Q3W) PLUS doxorubicin (A) 60 mg/m^2 in Cycles 6-9 on Day 1 (Q3W) PLUS cyclophosphamide (C) 600 mg/m^2 in Cycles 6-9 on Day 1 (Q3W). All treatments were administered via IV infusion except for doxorubicin (A), which was administered via IV injection. Each cycle was 21 days.
Arm/Group | Cohort A: KNp / KAC | Cohort B: KNpCb (Regimen 1) / KAC | Cohort C: KNpCb (Regimen 2) / KAC | Cohort D: KNpCb (Regimen 3) / KAC | Cohort E: KTCb (Regimen 1) / KAC | Cohort F: KTCb (Regimen 2) / KAC
All-Cause Mortality (participants affected / at risk) | 4/10 | 0/10 | 0/10 | 1/10 | 1/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 5/10 | 4/10 | 8/10 | 7/10 | 3/10 | 4/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 10/10 | 10/10 | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: KNp / KAC (N=10) | Cohort B: KNpCb (Regimen 1) / KAC (N=10) | Cohort C: KNpCb (Regimen 2) / KAC (N=10) | Cohort D: KNpCb (Regimen 3) / KAC (N=10) | Cohort E: KTCb (Regimen 1) / KAC (N=10) | Cohort F: KTCb (Regimen 2) / KAC (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 4 (4) | 4 (6) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subacute cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: KNp / KAC (N=10) | Cohort B: KNpCb (Regimen 1) / KAC (N=10) | Cohort C: KNpCb (Regimen 2) / KAC (N=10) | Cohort D: KNpCb (Regimen 3) / KAC (N=10) | Cohort E: KTCb (Regimen 1) / KAC (N=10) | Cohort F: KTCb (Regimen 2) / KAC (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 9 (14) | 7 (14) | 6 (7) | 7 (10) | 6 (13)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (6) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 4 (10) | 8 (24) | 7 (30) | 8 (25) | 4 (5) | 6 (7)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 7 (14) | 2 (4) | 4 (7) | 1 (1) | 2 (2)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (4) | 1 (2) | 1 (1) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (5) | 2 (3) | 2 (4) | 1 (2) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (4) | 4 (7) | 1 (1) | 5 (7) | 4 (7)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (9) | 4 (7) | 5 (7) | 3 (6)
Dyspepsia (Gastrointestinal disorders) | 4 (6) | 3 (6) | 1 (1) | 2 (3) | 4 (5) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (17) | 8 (22) | 10 (23) | 5 (13) | 8 (22) | 6 (9)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral mucosal blistering (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 2 (3) | 2 (5) | 4 (4) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (9) | 2 (3) | 4 (5) | 5 (11) | 4 (9) | 2 (4)
Asthenia (General disorders) | 3 (9) | 6 (8) | 3 (8) | 1 (1) | 2 (5) | 2 (3)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (7) | 3 (5) | 5 (12) | 3 (6) | 6 (6) | 6 (9)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal dryness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 6 (8)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Puncture site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Temperature regulation disorder (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspergillus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
External ear cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 3 (4) | 3 (3) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 2 (3) | 2 (4) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (4) | 1 (2) | 3 (3) | 2 (3) | 0 (0) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (2) | 2 (2) | 1 (2) | 0 (0) | 3 (3)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hepatic enzyme decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 2 (5) | 3 (5) | 2 (4) | 5 (11) | 2 (4)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 2 (3) | 1 (1)
Respirovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 2 (3) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 5 (6) | 4 (8) | 5 (7) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (2) | 3 (8) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Joint noise (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 4 (7) | 3 (6) | 0 (0) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 3 (4) | 5 (8) | 0 (0) | 2 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 3 (3)
Neurotoxicity (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5) | 1 (1) | 4 (6) | 2 (3) | 0 (0) | 2 (2)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Libido increased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulval ulceration (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (3) | 1 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4) | 5 (5) | 5 (5) | 5 (5) | 4 (4)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychalgia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (3) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (2) | 4 (6) | 5 (5) | 4 (5) | 2 (3)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vein disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Physical deconditioning (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT02622074/Prot_SAP_000.pdf